CLINICAL TRIAL: NCT02294708
Title: The Influence of Postoperative Postures on the Incidence and Duration of Persistent Sub-foveal Fluid After Scleral Buckle for Macula-off Retinal Detachment
Brief Title: The Influence of Postoperative Postures on Persistent Sub-foveal Fluid After Scleral Buckle Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Zhi-zhong Ma, chair of ophthalmology department, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PekingUTH-RD-2014
Record Dates: First submitted 2014-10-11; First posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Retinal Detachment
Keywords: macula-off retinal detachment; scleral buckle; persistent sub-foveal fluid; postoperative postures; optical coherence tomography (OCT)
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- supine (Experimental): postoperative postures: patients in this arm are assigned to adopt supine position for 24 hours after the surgery
  Interventions: Behavioral: postoperative postures
- temporal lateral (Experimental): postoperative postures: patients in this arm are assigned to adopt temporal lateral position for 24 hours after the surgery
  Interventions: Behavioral: postoperative postures

INTERVENTIONS:
Behavioral: postoperative postures — two postoperative postures: supine and temporal-lateral

SUMMARY:
The purpose of this study is to evaluate whether postoperative postures influence persistent sub-foveal fluid after scleral buckle surgery

DETAILED DESCRIPTION:
In this study, we are to compare the difference of influence of two postoperative postures on the incidence and duration of persistent sub-foveal fluid after scleral buckle surgery for macula-off retinal detachment

ELIGIBILITY:
Inclusion Criteria:

* rhegmatogenous retinal detachment (RRD)
* macula off
* treated by successful scleral buckle surgery
* recent onset with symptom within 1 month

Exclusion Criteria:

* with failed previous surgery
* intraoperative or postoperative injection of long-acting gas
* with other eye diseases than RRD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
duration of absorption of persistent sub-foveal fluid after surgery | Time from the date of operation until the date of absorption of sub-foveal fluid determined by OCT. The estimated period of time over which the event (absorption of sub-foveal fluid ) is assessed is up to 1 year.
  time interval from surgery to the date of disappearance of sub-foveal fluid on OCT

SECONDARY OUTCOMES:
best corrected visual acuity | 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Jin Chen, M.D., Study Director — Peking University Third Hospital; Chang-Guan Wang, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China